CLINICAL TRIAL: NCT06917794
Title: Development of Polygenic Risk Scores in Colon Cancer Patients Through the Study of Ancestry and Diversity in Genetic Maps of the Brazilian Population - ORIGEM Project
Acronym: ORIGEM
Status: Enrolling by invitation | Type: Observational
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Rodrigo Santa Cruz Guindalini, Doctor, D'Or Institute for Research and Education
Other Study IDs: 25000.130491/2023-48 - ORIGEM
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Colo-rectal Cancer; Polygenic Risk Score; Somatic Mutation; Hereditary Cancer; Germline Mutations; Cancer Predisposition Syndrome
MeSH Terms: conditions — Colonic Neoplasms; Genetic Risk Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Development of a polygenic risk score based on somatic and germline genetic information from patients with colorectal cancer

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer diagnosed in both men and women. Approximately 70% of CRC cases originate from spontaneous point mutations in oncogenes, tumor suppressor genes, and genes related to DNA repair mechanisms (Nigin et al., 2023). The remaining 30% result from hereditary mutations, of which 5-6% involve high-penetrance genes. Genetic predisposition due to pathogenic germline variants in high-risk cancer-associated genes has been implicated in 2-8% of all CRC cases, increasing to 6-10% when considering pathogenic mutations in both high- and moderate-penetrance genes.

For individuals with certain hereditary cancer syndromes, the risk of developing colorectal cancer can reach 50-80% in the absence of endoscopic and/or surgical intervention. Therefore, characterizing high-, moderate-, and low-penetrance genes within a population is crucial for understanding hereditary tumorigenesis and guiding more cost-effective screening strategies.

Genetic studies comparing genomes from populations of different ethnic backgrounds have demonstrated that ancestry plays a significant role in genetic predisposition to CRC. Given the high level of genetic admixture in the Brazilian population, studies focused solely on populations of European ancestry fail to provide a representative model for application in highly admixed populations like Brazil.

In this context, the present study aims to utilize next-generation sequencing (NGS) in a cohort representative of the Brazilian population with CRC and controls to develop a Polygenic Risk Score (PRS). This score could impact cancer screening and prevention strategies, as well as genetic counseling for patients and their families. The hypothesis is that genetic mapping-including ancestry, germline, and tumor genetic variability-in Brazilian colorectal cancer patients will provide valuable data for developing a PRS that may eventually guide more targeted and cost-effective screening strategies for our population.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years;
* Histologically confirmed diagnosis of colorectal cancer;
* Have available tumor material for somatic sequencing, obtained from biopsy or routine surgery;
* Sign the informed consent form (ICF) for the study.

Exclusion Criteria:

• Pregnants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Of the 500 patients included, approximately 56% will be recruited from participants self-identified as brown, black, or indigenous, with the remaining percentage distributed between white and yellow. Of these individuals, at least 50% will be women, corresponding to the sex and race distribution in the Brazilian population reported in the latest IBGE census in 2022.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Elaboration of Poligenic Risk | 36mo
  A germline and somatic genetic mapping in Brazilian patients with colon adenocarcinoma, including ancestry, for the development of a polygenic risk score system applicable to the Brazilian population.

CONTACTS AND LOCATIONS:
Locations (9):
- Brazil (9):
  - Instituto D'Or de Pesquisa e Ensino, Fortaleza, Ceará
  - CPOC - Centro de Pesquisa Oncológica e Clínica, faz parte do Complexo Associação Obras Sociais lrmã Dulce (AOSID), Salvador, Estado de Bahia
  - Instituto D'Or de Pesquisa e Ensino, Salvador, Estado de Bahia
  - Instituto D'Or de Pesquisa e Ensino, Brasília, Federal District
  - Instituto D'Or de Pesquisa e Ensino, Curitiba, Paraná
  - Instituto D'Or de Pesquisa e Ensino, Recife, Pernambuco
  - Instituto D'Or de Pesquisa e Ensino, Rio de Janeiro, Rio de Janeiro
  - Instituto D'Or de Pesquisa e Ensino, São Paulo, São Paulo
  - Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No